CLINICAL TRIAL: NCT02923427
Title: Comparison of I-gel and LMA Supreme Without Neuromuscular Blocker in Laparoscopic Gynecological Surgery
Brief Title: I-gel vs LMA Supreme in Laparoscopic Gynecological Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Sule Ozbilgin, Dokuz Eylul University, MD, Anesthesiologists., Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 266-SBKAEK
Record Dates: First submitted 2016-09-22; First posted 2016-10-04 (Estimated); Results first posted 2020-10-08 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Airway Morbidity; Anaesthesia
Keywords: laryngeal mask Supreme; i-gel; laparoscopic gynecological surgery

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Laryngeal mask Supreme (Active Comparator): Insertion of the "Laryngeal mask Supreme" and evaluation of its clinical performance
  Interventions: Device: Laryngeal mask Supreme Evaluation
- i-gel (Experimental): Insertion of the "i-gel" and evaluation of its clinical performance
  Interventions: Device: i-gel Evaluation

INTERVENTIONS:
Device: Laryngeal mask Supreme Evaluation — Evaluation of clinical performance in terms of Insertion, ventilation and complications
  Arms: Laryngeal mask Supreme
Device: i-gel Evaluation — Evaluation of clinical performance in terms of Insertion,ventilation and complications
  Arms: i-gel

SUMMARY:
To compare the effects of i-gel and Laryngeal mask airway Supreme (LMA-Supreme) on ventilation parameters and surgical view during Trendelenburg Position laparoscopic gynecological surgery in cases administered positive pressure ventilation without the use of neuromuscular agents.

DETAILED DESCRIPTION:
Prospective, randomized and double-blind study, aged from 18 to 65 years undergoing elective laparoscopic gynecological surgery.

The patients are randomly assigned to 2 groups:

* Group 1: i-gel
* Group 2: LMA- Supreme

Procedure:

The investigation protocol contains the following sections:

1. Induction of anaesthesia. For preoperative sedation 0.02 mg/kg midazolam IV will be administered. 2 minutes of 0.2 µ/kg/min remifentanil and 6 mg kg st-1 propofol infusion, IV 1-2 mg kg-1 propofol . No muscle relaxant will be used for insertion of the airway device.
2. Bispectral index values will be held between 40-60.Bispectral index values will be within this interval by increasing or decreasing propofol infusion by 1 mg/kg after additional bolus dose of propofol (1 mg/kg).
3. Insertion of the airway device. The size of the airway device used is based on the manufacturers' recommendations. All devices are deflated a lubricated prior to use. Once inserted, the cuff is be inflated with a manometer up to 60 cm H20 Data recorded: size of airway device, time an number of attempts.
4. Anesthesia maintenance will be ensured by 50% O2/air with 0.1-0.4 µ kg/min-1 remifentanil and 50-150 µ kg/ min-1 (4-10 mg/kg/hr) propofol IV infusion
5. Functionality of the gastric drainage channel of the airway device: passage of a 14 G size tube.
6. Measurement of airway seal pressure (oropharyngeal leak pressure (OLP): at baseline, and at 2 minutes after airway device insertion (T1), 10 minutes after insufflation (T2), before desufflation (T3), before removal of airway device (T4). The maximum pressure allowed is 40 cm H2O.
7. Ventilatory mechanics and parameters and hemodynamic parameters are measured at baseline, and at T1, T2, T3 and T4.
8. Perioperative complications: Cough, vomiting, laryngeal spasm, laryngeal Stridor, airway intervention requirements, hypoxia (SpO2 < 92%)
9. Removal of the airway device: Presence of blood - 3 level grading (1:no blood; 2: trace amounts of blood; 3: clear amounts of blood). Complications: sore throat ( VAS:10-point scale), dysphonia (yes/no), dysphagia (yes/no).

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesiologists classification group I-II
2. between 18-65 years
3. undergoing elective laparoscopic gynecological surgery

Exclusion Criteria:

1. Those with any neck or upper respiratory tract pathology
2. Those at risk of gastric content regurgitation/aspiration (previous upper Gastrointestinal system surgery, known hiatus hernia, gastroesophageal reflux, history of peptic ulcers, full stomach, pregnancy)
3. Those with low pulmonary compliance or high airway resistance (chronic pulmonary diseases)
4. Obese patients (BMI >35)
5. Those with throat pain, dysphagia and dysphonia
6. Those with possible or previous difficult airway
7. Those with operations planned for longer than 4 hours
8. Conversion to laparatomy
9. Neuromuscular blocking agent used

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ferim Günenç, MD, Study Director — Dokuz Eylül University, School of Medicine, Department of Anesthesiology and Reanimation
Locations (1):
- Dokuz Eylül University, School of Medicine, Department of Anesthesiology and Reanimation, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Laryngeal Mask Supreme | I-gel
Started | 55 | 57
Completed | 51 (The reasons: n= 2 Convert to Laparotomy n=1 Desaturation n=1 LMA-S can not be placed) | 55 (The reasons: n = 2 Convert to Laparotomy)
Not Completed | 4 | 2
Not completed — convert to laparatomy | 2 | 2
Not completed — destaturation | 1 | 0
Not completed — can not replace LMA | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Laryngeal Mask Supreme | I-gel | Total
Number analyzed (Participants) | 51 | 55 | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.55 (9.34) | 36.44 (8.31) | 35.49 (8.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 55 | 106
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Turkey | 51 | 55 | 106

OUTCOME MEASURES:

1. Primary Outcome: Airway Seal Pressure Values
Description: This value is important as it indicates the feasibility of positive pressure ventilation and the degree of airway protection from supracuff soiling. It is also used in LMA studies as an index of successful placement.Airway pressures of ≈20 cm H2O are typically required in routine practice.
Time Frame: At baseline and at 15, 30 and 60 minutes
Measure: Mean (Standard Deviation); unit: cm H2O
Arm/Group | Laryngeal Mask Supreme | I-gel
Number analyzed (Participants) | 51 | 55
cm H2O
  baseline | 31.20 (8.07) | 27.58 (7.16)
  at 15 min | 30.10 (6.48) | 28.76 (7.33)
  at 30 min | 29.92 (6.19) | 28.71 (6.65)
  at 60 min | 30.31 (6.19) | 29.13 (6.47)

2. Secondary Outcome: Visual Quality
Description: quality of surgical view will evaluate by the scala. quality of surgical view will be assessed with points from 1 to 4 by the surgeon blind to the airway device; (1:best, 4: worst).
Time Frame: during pneumoperitoneum
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Laryngeal Mask Supreme | I-gel
Number analyzed (Participants) | 51 | 55
units on a scale | 3.941 (0.42) | 3.945 (0.40)

3. Secondary Outcome: Gastric Tube Insertion
Description: Number of Participants According to Ease of Gastric Tube Insertion.Ease of passage of a gastric tube as: very easy, easy, difficult or very difficult.
Time Frame: following airway device insertion up to 5 minutes
Measure: Number; unit: participants
Arm/Group | Laryngeal Mask Supreme | I-gel
Number analyzed (Participants) | 51 | 55
participants
  very easy | 33 | 12
  easy | 18 | 27
  difficult | 0 | 10
  very difficult | 0 | 6

4. Secondary Outcome: Postoperative Pharyngolaryngeal Morbidity
Description: Sore throat evaluted by Visual Analogue Scale. The visual analog scale, also known as the graphic rating scale is a simple, valid and reliable subjective measure. Scores are ranked on a 10-cm line that stretches between two extremes - "no pain" and "worst pain". Total range provided"0 (no pain) to 10 (worst pain).
Time Frame: postoperative first hour and 24th hour
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Laryngeal Mask Supreme | I-gel
Number analyzed (Participants) | 51 | 55
units on a scale
  at first hour | 0.43 (1.02) | 0.16 (0.06)
  24th hour | 0.02 (0.140) | 0.00 (0.00)

5. Secondary Outcome: Sufficiency of Pneumoperitoneum
Description: Number of Participants with Sufficiency of Pneumoperitoneum. Sufficiency of pneumoperitoneum for the surgical procedure according to surgeon, described as sufficient or insufficient questionaire.
Time Frame: baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Laryngeal Mask Supreme | I-gel
Number analyzed (Participants) | 51 | 55
Participants
  sufficient | 50 | 55
  insufficient | 1 | 0

6. Secondary Outcome: Mean Airway Pressure Values
Description: Mean airway pressure typically refers to the mean pressure applied during positive-pressure mechanical ventilation. Mean airway pressure correlates with alveolar ventilation, arterial oxygenation, hemodynamic performance, and barotrauma.
Time Frame: At baseline and at 15, 30 and 60 minutes
Measure: Mean (Standard Deviation); unit: cm H2O
Arm/Group | Laryngeal Mask Supreme | I-gel
Number analyzed (Participants) | 51 | 55
cm H2O
  baseline | 5.84 (0.92) | 5.82 (1.09)
  at 15 min | 7.84 (1.23) | 7.87 (1.47)
  at 30 min | 7.45 (1.31) | 7.27 (1.39)
  at 60 min | 6.51 (1.15) | 6.29 (1.21)

7. Secondary Outcome: Dysphonia With Yes/no.
Description: We evaluated while a patient was talking with us that the patient has dysphonia or not .
Time Frame: postoperative first hour and 24th hour
Measure: Number; unit: Number of Participants without Dysphonia
Arm/Group | Laryngeal Mask Supreme | I-gel
Number analyzed (Participants) | 51 | 55
Number of Participants without Dysphonia
  at first hour-no | 51 | 55
  at 24th hour-no | 51 | 55

8. Secondary Outcome: Disphagia
Description: We asked the question that you have a pain while you were swallowing, yes or not.
Time Frame: postoperative first hour and 24th hour
Measure: Count of Participants; unit: Participants
Arm/Group | Laryngeal Mask Supreme | I-gel
Number analyzed (Participants) | 51 | 55
Participants
  at first hour-no | 47 | 54
  at 24th hour-no | 51 | 55

ADVERSE EVENTS:
Time Frame: 24 hour
Arm/Group | Laryngeal Mask Supreme | I-gel
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/55
Other Adverse Events (participants affected / at risk) | 0/51 | 0/55

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-21): https://cdn.clinicaltrials.gov/large-docs/27/NCT02923427/Prot_SAP_000.pdf